CLINICAL TRIAL: NCT04126746
Title: Clinical Trials in Organ Transplantation Extension Study (CTOT-ES)
Brief Title: Clinical Trials in Organ Transplantation Extension Study
Acronym: CTOT-ES
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00102592; PALMER19AB0 (Other Grant/Funding Number: Cystic Fibrosis Foundation)
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Lung Transplant Failure and Rejection
Keywords: Lung transplantation; Chronic lung allograft dysfunction
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Bronchoaveolar lavage fluid - lung fluid obtained during a bronchoscopy procedure
  Blood collection by needle stick; blood collection separated into its components of serum, plasma, RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to continue to follow subjects who were enrolled in the CTOT-20 CLAD Phenotypes study. Subjects will provide clinical data and complete quality of life questionnaires that will be used to determine the clinical factors associated with the development of Chronic Lung Allograft Dysfunction (CLAD) after lung transplant.

DETAILED DESCRIPTION:
There are no mandated study visits, rather the study will be conducted using real world data collected as part of usual clinical care according to the standard of care transplant protocols at each site. Specimens and study data will be collected during standard of care visits and study coordinators will review medical records and extract available clinical data every 6 months. Study coordinators will collect Pulmonary Function Test data that will be transferred to the Data Coordinating Center as in CTOT-20. Subjects will be asked to complete quality of life questionnaires on an annual basis.

The majority of times, blood samples will be collected during clinical care routine venipuncture based on clinic visit scheduling. In the rare circumstances in which research blood is missed during a standard of care venipuncture or one is not scheduled, a participant may be asked to undergo venipuncture for study purposes.

Standard of care (SOC) bronchoscopies with collection of Bronchoalveolar Lavage (BAL) lung fluid will be performed at each center according to clinical management protocols. During SOC bronchoscopies, research participants will undergo additional fluid instillation for research BAL sampling as in CTOT-20.

ELIGIBILITY:
Inclusion Criteria:

* Current CTOT-20 participants

Exclusion Criteria:

* Non-CTOT-20 participants
* Withdrawn CTOT-20 participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include participants previously enrolled in the CTOT-20 study who are alive and remain active in the study (i.e. not previously withdrawn). The CTOT-20 cohort consists of adults who received their first lung transplant at one of the five participating centers (Duke University Medical Center, University of California Los Angeles Medical Center, Cleveland Clinic Foundation, Johns Hopkins University, Toronto General Hospital). Multi-organ recipients as well as prior recipients of any solid organ or bone marrow transplant were excluded. Recipients with HIV infection were excluded as were those participating in an investigational drug trial at the time of enrollment. At the time of this protocol writing, there are 625 out of 803 CTOT-20 participants alive and active in follow-up, who are eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Time from lung transplant to Chronic Lung Allograft Dysfunction (CLAD) (including RCLAD or BOS) as measured by serial pulmonary function tests | Baseline, up to 24 months
  Time from lung transplant to the development of CLAD (Restrictive Chronic Lung Allograft Dysfunction (RCLAD) or Bronchiolitis Obliterans Syndrome (BOS) as measured by a change in pulmonary function and Physician Adjudication
Number of participants that develop CLAD as measured by change in pulmonary function and Physician Adjudication | Up to 24 months
Number of participants that have Th1, Th2, Th17 immune profiles as measured in the lung fluid | Up to 24 months
Number of participants that have Th1, Th2, and Th17 immune profiles as measured in the blood | Up to 24 months

SECONDARY OUTCOMES:
Change in Quality of Life (QOL) as serially assessed by the Short Form 36 (SF-36) | Baseline and annually for 2 years
  The SF-36 is a 36 item survey that measures personal views on health and activities of daily living.
Change in Quality of Life (QOL) as serially assessed by the Saint George's Respiratory Questionnaire | Baseline and annually for 2 years
  The Saint George's Respiratory Questionnaire is a 2 part questionnaire that measures troubled breathing and the impact on quality of life.
Time from CLAD onset to death as measured by medical record review | Up to 24 months
Time from CLAD onset to retransplant as measured by medical record review | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Palmer, MD, MHS, Principal Investigator — Duke University
Locations (5):
- United States (4):
  - University of California Los Angeles Medical Center, Los Angeles, California
  - Johns Hopkins University, Baltimore, Maryland
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No